CLINICAL TRIAL: NCT05285306
Title: Developing and Pilot Testing a Brief Intervention to Reduce Anxiety During Pelvic Examinations Among Female Cancer Survivors (Pelvic Examination and Anxiety Coping Skills for Empowerment: PEACE)
Brief Title: Surveillance Pelvic Examination Anxiety: Brief Coping Skills Intervention
Acronym: PEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00107843
Record Dates: First submitted 2022-03-07; First posted 2022-03-17 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2021-11

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEACE Program (Experimental): 3 sessions of tailored coping skills related to pelvic examinations
  Interventions: Behavioral: PEACE Program

INTERVENTIONS:
Behavioral: PEACE Program — This pilot will consist of 3 individual telemedicine sessions to teach cognitive behavioral coping skills and provide education related to gynecologic cancer surveillance and psychological distress.
  Other Names: Pelvic Exam and Anxiety Coping Skills for Empowerment

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of a brief coping skills training program addressing anxiety and pain related to surveillance pelvic examinations for female gynecologic cancer survivors.

DETAILED DESCRIPTION:
The investigators have developed and manualized a coping skills training intervention for female gynecologic cancer patients that aims to reduce anxiety related to surveillance pelvic examinations (Pelvic Examination and Anxiety Coping Skills for Empowerment: PEACE). The investigators propose a proof-of concept pilot study to evaluate the acceptability and feasibility of the coping skills intervention. The study will be conducted by Duke University. Participants (N=16) will receive the 3-session telemedicine coping skills intervention. Participants will complete assessments at baseline, post-intervention (within 2 weeks before their next scheduled pelvic examination), and post pelvic examination (2-3 months after the baseline assessment). Study aims are: Aim 1) Assess intervention acceptability and feasibility through quantitative measurement and qualitative feedback from semi-structured interviews, and Aim 2) Graphically depict patterns of change in outcome variables and intervention targets.

ELIGIBILITY:
Inclusion Criteria:

* female sex
* diagnosis of stage I-IV cervical or endometrial cancer
* 18 years of age or older
* able to speak/read English
* able to give informed consent
* completed cancer treatments within 2-24 months prior to enrollment, and recommended to undergo surveillance pelvic examination at three month intervals
* able to commit to three 45-60 minute visits within the study period
* able to participate in the intervention via the telemedicine modality (e.g., phone or video)

Exclusion Criteria:

* unable to provide informed consent
* major untreated or uncontrolled mental illness
* hearing impairment that impedes telephone or video calls

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 16 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Intervention acceptability will be assessed using an adapted version of the Satisfaction with Therapy and Therapist Scale (STTS-R) | post pelvic examination (approximately 2-3 months after baseline)
  The adapted STTS-R consists of 18 items that assess satisfaction with the therapist and the intervention on a 5-point Likert-type scale from 1 (strongly disagree) to 5 (strongly agree).
Change in intervention acceptability will be assessed using an adapted version of the Satisfaction with Therapy and Therapist Scale (STTS-R) | post-intervention (within 2 weeks of their next pelvic examination), post pelvic examination (approximately 2-3 months after baseline)
  Change in intervention acceptability from immediately after completion of the 3 sessions (post intervention assessment) to after trying to implement the coping skills during their next pelvic examination (post pelvic exam assessment), using the STTS-R. The adapted STTS-R consists of 18 items that assess satisfaction with the therapist and the intervention on a 5-point Likert-type scale from 1 (strongly disagree) to 5 (strongly agree).
Intervention feasibility as measured by percentage of recruited participants who enrolled | post pelvic examination (approximately 2-3 months after baseline)
  Enrollment logs will capture the number of participants who were recruited and among them, the number that enrolled in the study.
Intervention feasibility as measured by attrition | post pelvic examination (approximately 2-3 months after baseline)
  Retention logs will capture the number of participants who did not complete the study protocol (rate of attrition)
Intervention feasibility as measured by survey completion | post pelvic examination (approximately 2-3 months after baseline)
  Retention logs will capture the number of participants who completed all assessments
Intervention feasibility as measured by home practice completion | post-intervention (within 2 weeks of their next pelvic examination)
  Interventionist logs completed at the conclusion of each session will capture the level of home practice completion
Intervention feasibility as measured by participant engagement | post-intervention (within 2 weeks of their next pelvic examination)
  Interventionist logs completed at the conclusion of each session will capture the level of participant engagement with a 1 item question rated from 1 (not at all engaged) to 4 (highly engaged).
Intervention feasibility as measured by interventionist fidelity | post-intervention (within 2 weeks of their next pelvic examination)
  Fidelity rating forms will be used to measure the level of fidelity to session content for one third of the sessions for the protocol. Each component of the session will be rated from 0 (not covered at all) to 3 (thoroughly covered the topic)

SECONDARY OUTCOMES:
Change in anxiety related to examination as measured by the The State Anxiety Scale of the State-Trait Anxiety Inventory | baseline, post-intervention (within 2 weeks of their next pelvic examination), post pelvic examination (approximately 2-3 months after baseline)
  The State Anxiety Scale of the STAI is comprised of 20 items on a 5-point Likert scale, which range from 1 (not at all) through 4 (very much).
Change in pain during examination as measured by numeric scales | baseline, post pelvic examination (approximately 2-3 months after baseline)
  Numeric scales will be used to assess the average pain during examination, worst pain during examination, and lowest pain during examination, ranging from 0 (no pain) to 10 (pain as bad as you could imagine). The three pain intensity ratings will be averaged to create a total score for pain.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Shelby, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No